CLINICAL TRIAL: NCT02085980
Title: Clinical Investigation to Assess the Safety and Efficacy of the Laser for the Treatment of Vulvovaginal Atrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: El. En. SpA (Industry)
Collaborators: The Christ Hospital (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELEN13-VVA-MK01
Record Dates: First submitted 2014-03-10; First posted 2014-03-13 (Estimated); Results first posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2017-02

CONDITIONS: Vulvovaginal Atrophy
MeSH Terms: interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laser Treatment (Experimental): Laser Treatment
  Interventions: Device: Laser treatment

INTERVENTIONS:
Device: Laser treatment — The laser handpiece (probe) will be deposited in the vaginal canal and the laser energy will be delivered through the handpiece

SUMMARY:
The purpose of this study is to assess the safety and the efficacy of a laser in the treatment of vulvovaginal atrophy (VVA), that is to assess the change in the severity of the vaginal dryness symptom, by means of a visual analogic scale (10 cm VAS).

DETAILED DESCRIPTION:
The laser handpiece (probe) will be deposited in the vaginal canal and the laser energy will be delivered through the handpiece. Subjects will receive a total of three (3) treatments every six (6) weeks (+/-1 week). Subjects will return one week (+/- 3 days) post the first treatment, as well as three (3) months (+/- 2 weeks) and twelve (12) months (+/- 2 weeks) post the third treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smoking post menopausal women with absence of menstruation of at least 12 months
* Exhibiting VVA symptoms
* Prolapse staged < II, according to the pelvic organ prolapse quantification (ICS-POP-Q) system
* Have not had procedures in the anatomical area through 6 months prior to treatment
* Understand and accept the obligation and is logistically able to present for all scheduled follow-up visits

Exclusion Criteria:

* • Acute or recurrent urinary tract infection (UTI), or genital infection (e.g. herpes candida).

  * Prolapse staged ≥ II, according to the pelvic organ prolapse quantification (ICS-POP-Q) system
  * Any serious disease, or chronic condition, that could interfere with the study compliance
  * Previously undergone reconstructive pelvic surgery
  * Have used vaginal creams, moisturizers, lubricants or homeopathic preparations for at least 3 months
  * A history of thrombophlebitis
  * A history of acute infections
  * A history of heart failure
  * Received or is anticipated to receive antiplatelets, anticoagulants, thrombolytics, vitamin E or anti inflammatories within 2 weeks pre treatment
  * Any medical condition, that, in the investigator's opinion would interfere with the patient's participation in the study
  * Taking medications that are photosensitive
  * A history of keloid formation

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mickey Karram, MK, Principal Investigator — Hospital Physician, The Christ Hospital; Eric Sokol, MD, Study Director — Stanford University
Locations (2):
- United States (2):
  - Stanford University, Palo Alto, California
  - The Carl and Edyth Lindner Center for Research and Education at The Christ Hospital, West Chester, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] van der Laak JA, de Bie LM, de Leeuw H, de Wilde PC, Hanselaar AG. The effect of Replens on vaginal cytology in the treatment of postmenopausal atrophy: cytomorphology versus computerised cytometry. J Clin Pathol. 2002 Jun;55(6):446-51. doi: 10.1136/jcp.55.6.446. PMID 12037029

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Laser Treatment
Started | 30
Completed | 27
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Laser Treatment
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: The Main Outcome of the Study is the Efficacy of the Laser Procedure, Intended as the Amelioration of 50% of the Severity of the Vaginal Dryness at 12 Months, Compared With Baseline
Description: The main outcome of the study is the efficacy of the laser procedure, intended as the amelioration of 50% of the severity of the vaginal dryness at 12 months, compared with baseline.
  The change in the vaginal dryness symptom has been assessed by means of a visual analogic scale (10 cm VAS).
Time Frame: Baseline and at follow up visit at 12 months post last treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Laser Treatment
Number analyzed (Participants) | 30
Participants | 27

ADVERSE EVENTS:
Arm/Group | Laser Treatment
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No